CLINICAL TRIAL: NCT00796445
Title: GSK 2132231A Antigen-Specific Cancer Immunotherapeutic as Adjuvant Therapy in Patients With Resected Melanoma
Brief Title: A Phase III Study to Test the Benefit of a New Kind of Anti-cancer Treatment in Patients With Melanoma, After Surgical Removal of Their Tumor
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early following assessment of the two co-primary endpoints showing the lack of efficacy of the study product.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111482; 2008-002447-16 (EudraCT Number)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
Keywords: DERMA; Tumor antigen; Immunotherapeutic; Adjuvant cancer therapy; Melanoma; ASCI
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- MAGE-A3 Group (Experimental): Patients who received up to 13 doses of recMAGE-A3 + AS15 ASCI. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of ASCI product at 3-week intervals, followed by 8 doses of ASCI product at 12-week intervals.
  Interventions: Drug: GSK 2132231A
- Placebo Group (Placebo Comparator): Patients who received up to 13 doses of placebo. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of placebo at 3-week intervals, followed by 8 doses of placebo at 12-week intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK 2132231A — IM solution, a course of 13 injections administered over 27 months
  Arms: MAGE-A3 Group
Drug: Placebo — IM solution, a course of 13 injections administered over 27 months
  Arms: Placebo Group

SUMMARY:
The purpose of this clinical trial is to evaluate the benefit of the immunotherapeutic product GSK 2132231A in preventing disease relapse when given to melanoma patients, after surgical removal of their tumor.

This Protocol Posting has been updated following Amendments 1 of the Protocol, March 2010. The impacted sections are outcome measures and entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed.
* Male or female patient with histologically proven stage IIIB or IIIC cutaneous melanoma presenting with macroscopic lymph node involvement suitable for surgery.
* The patient must have been surgically rendered free of disease before the randomization.
* Patient is ≥ 18 years old at the time of signing the informed consent form.
* The patient's lymph node tumor shows expression of the MAGE-A3 gene.
* The patient has fully recovered from surgery.
* ECOG performance status of 0 or 1 at the time of randomization.
* The patient must have adequate organ functions as assessed by standard laboratory criteria.
* If the patient is female, she must be of non-childbearing potential, or practice adequate contraception.
* In the opinion of the investigator, the patient can and will comply with all the requirements of the protocol.

Exclusion Criteria:

* The patient suffers from a mucosal or ocular melanoma.
* The patient has or has had any history of in-transit metastases
* The patient has been treated or is scheduled to be treated with an adjuvant anticancer therapy after the surgery that qualifies the patient for inclusion in the present trial.
* The patient requires concomitant chronic treatment with systemic corticosteroids or any other immunosuppressive agents.
* Use of any investigational or non-registered product (drug or vaccine) other than the study treatment.
* The patient has a history of autoimmune disease.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient is known to be positive for Human Immunodeficiency Virus (HIV) or has another confirmed or suspected immunosuppressive or immunodeficient condition.
* History of allergic disease or reactions likely to be exacerbated by any component of the treatments.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
* The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* The patient has an uncontrolled bleeding disorder.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (225):
- United States (62):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orange Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Latham, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sayre, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (4):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Cipolletti, Río Negro Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Australia (9):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, North Sydney, New South Wales
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Brisbane, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
- Austria (6):
  - GSK Investigational Site, Feldkirch
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Wels
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Wilrijk
- Brazil (3):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Canada (2):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ottawa, Ontario
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (23):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Boulogne
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Villejuif
- Germany (34):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Buxtehude, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Oldenburg, Lower Saxony
  - GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Quedlinburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
- GSK Investigational Site, Athens, Greece
- Ireland (3):
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
- Israel (3):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
- Italy (11):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Aviano (PN), Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Padua, Veneto
- Japan (2):
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Monterrey, Nuevo León, Mexico
- Netherlands (2):
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Wellington
- GSK Investigational Site, Oslo, Norway
- Poland (7):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Warsaw
- Romania (3):
  - GSK Investigational Site, Baia Mare
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova, Dolj
- Russia (6):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Stavropol
- Serbia (2):
  - GSK Investigational Site, Belgrade
  - GSK Investigational Site, Kamenitz
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Uppsala
- Switzerland (2):
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Zurich
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien
- Ukraine (5):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kryvyi Rih
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
- United Kingdom (7):
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Belfast, Northern Ireland
  - GSK Investigational Site, Colchester
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, London
  - GSK Investigational Site, Poole, Dorset
  - GSK Investigational Site, Salisbury

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=16038

REFERENCES:
- [Background] Dreno B, Thompson JF, Smithers BM, Santinami M, Jouary T, Gutzmer R, Levchenko E, Rutkowski P, Grob JJ, Korovin S, Drucis K, Grange F, Machet L, Hersey P, Krajsova I, Testori A, Conry R, Guillot B, Kruit WHJ, Demidov L, Thompson JA, Bondarenko I, Jaroszek J, Puig S, Cinat G, Hauschild A, Goeman JJ, van Houwelingen HC, Ulloa-Montoya F, Callegaro A, Dizier B, Spiessens B, Debois M, Brichard VG, Louahed J, Therasse P, Debruyne C, Kirkwood JM. MAGE-A3 immunotherapeutic as adjuvant therapy for patients with resected, MAGE-A3-positive, stage III melanoma (DERMA): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Jul;19(7):916-929. doi: 10.1016/S1470-2045(18)30254-7. Epub 2018 Jun 13. PMID 29908991
- [Background] Dizier B, Callegaro A, Debois M, Dreno B, Hersey P, Gogas HJ, Kirkwood JM, Vansteenkiste JF, Sequist LV, Atanackovic D, Goeman J, van Houwelingen H, Salceda S, Wang F, Therasse P, Debruyne C, Spiessens B, Brichard VG, Louahed J, Ulloa-Montoya F. A Th1/IFNgamma Gene Signature Is Prognostic in the Adjuvant Setting of Resectable High-Risk Melanoma but Not in Non-Small Cell Lung Cancer. Clin Cancer Res. 2020 Apr 1;26(7):1725-1735. doi: 10.1158/1078-0432.CCR-18-3717. Epub 2019 Nov 15. PMID 31732522
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 1351 patients enrolled in the study, 6 patients did not receive treatment and were excluded from study start, hence 1345 patients were included in the Total treated population-as treated (895 in the MAGE-A3 Group and 450 in the Placebo Group). Between the final and follow-up analyses, 1 patient was found to have an invalid ICF and was not included in the follow-up analysis, which included 1344 patients: 894 in the MAGE-A3 Group and 450 in the Placebo Group.
Period: Overall Study
Arm/Group | MAGE-A3 Group | Placebo Group
Started | 895 | 450
Completed | 310 | 158
Not Completed | 585 | 292
Not completed — Protocol Violation | 5 | 3
Not completed — Adverse event, serious fatal | 10 | 5
Not completed — Adverse event, non-fatal | 4 | 0
Not completed — Disease progression/recurrence | 537 | 268
Not completed — Other | 10 | 7
Not completed — Withdrawal by Subject | 18 | 9
Not completed — Invalid Informed Consent Form | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MAGE-A3 Group: Patients who received up to 13 doses of recMAGE-A3 + AS15 ASCIStudy products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of ASCI product at 3-week intervals, followed by 8 doses of ASCI product at 12-week intervals.
- Total: Total of all reporting groups
Arm/Group | MAGE-A3 Group | Placebo Group | Total
Number analyzed (Participants) | 895 | 450 | 1345
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (13.51) | 56.2 (13.66) | 56.1 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 345 | 188 | 533
  Male | 550 | 262 | 812
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian - Japanese Heritage | 4 | 3 | 7
  Geographic ancestry: White - Arabic/North African Heritage | 4 | 1 | 5
  Geographic ancestry: White - Caucasian/European Heritage | 880 | 443 | 1323
  Geographic ancestry: Other - Mixed origin | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: DFS = time to event from randomization to the date of first disease recurrence (as assessed by investigator) or the date of death (whatever cause), whichever occurred first. DFS was expressed as the person-year rate i.e. the number of patients with at least one event (n) over the sum of the follow-up periods in years (T), until the first occurrence of a recurrence/death. Types of recurrence to be considered as an event included loco-regional and distant metastases. Any death occurring without prior documentation of tumor recurrence was considered as an event (not censored in the stat. analysis) as this approach was less prone to introduce bias. If no event occurred by the time of analysis, then the time to event was censored at the last assessment date (tumor assessment/visit) of the patient. Any new primary cancer at another site, including second primary melanoma, was not considered as a recurrence and had to be reported as a Serious Adverse Event (SAE).
Time Frame: At Final analysis (Month 30 = Year 2.5)
Population: The analysis was performed on the Total Treated population - as randomized, which included patients in the treatment groups as allocated by the randomization system at the start of the study.
Measure: Number; unit: First events per person-year
Groups:
- GS+ Mage-A3 Sub-Group: Subset of patients with the pre-specified gene signature (GS+), receiving the MAGE-A3 ASCI product. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of ASCI product at 3-week intervals, followed by 8 doses of ASCI product at 12-week intervals.
- GS+ Placebo Sub-Group: Subset of patients with the pre-specified gene signature, receiving placebo. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of placebo at 3-week intervals, followed by 8 doses of placebo at 12-week intervals.
- GS- Mage-A3 Sub-Group: Subset of patients without the pre-specified gene signature (GS-), receiving the MAGE-A3 ASCI product. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of ASCI product at 3-week intervals, followed by 8 doses of ASCI product at 12-week intervals.
- GS- Placebo Sub-Group: Subset of patients without the pre-specified gene signature, receiving placebo. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of placebo at 3-week intervals, followed by 8 doses of placebo at 12-week intervals.
Arm/Group | MAGE-A3 Group | Placebo Group | GS+ Mage-A3 Sub-Group | GS+ Placebo Sub-Group | GS- Mage-A3 Sub-Group | GS- Placebo Sub-Group
Number analyzed (Participants) | 893 | 452 | 200 | 116 | 255 | 126
First events per person-year | 0.505 | 0.478 | 0.500 | 0.460 | 0.437 | 0.442
Statistical Analysis 1: Comparison: MAGE-A3 Group vs Placebo Group; At Final analysis (Month 30); Test type: Non-Inferiority — The aim of this analysis was to demonstrate the clinical efficacy in terms of disease-free survival (DFS) of recMAGE-A3 + AS15 ASCI compared to placebo in the overall study population of patients with completely resected stage III cutaneous melanoma with macroscopic lymph node involvement; p = 0.8566, Regression, Cox; Hazard Ratio (HR) = 1.013, 95% CI 2-sided [0.879 to 1.169]
Statistical Analysis 2: Comparison: GS+ Mage-A3 Sub-Group vs GS+ Placebo Sub-Group; At Final analysis (Month 30); Test type: Non-Inferiority — The aim of this analysis was to demonstrate the clinical efficacy in terms of DFS of the recMAGE-A3 + AS15 ASCI compared to placebo in the population presenting the potentially favorable gene expression signature; p = 0.4821, Regression, Cox; Hazard Ratio (HR) = 1.111, 95% CI 2-sided [0.828 to 1.491]
Statistical Analysis 3: Comparison: GS- Mage-A3 Sub-Group vs GS- Placebo Sub-Group; At Final analysis (Month 30); Test type: Non-Inferiority — The aim of this analysis was to demonstrate the clinical efficacy in terms of DFS of the recMAGE-A3 + AS15 ASCI compared to placebo in the population without the potentially favorable gene expression signature; p = 0.5375, Regression, Cox; Hazard Ratio (HR) = 0.915, 95% CI 2-sided [0.691 to 1.212]

2. Primary Outcome: Disease Free Survival (DFS)
Description: as for outcome 1
Time Frame: At follow-up analysis (up to Year 5)
Population: The analysis was performed on the Total Treated population - as randomized, which included patients in the treatment groups as allocated by the randomization system at the start of the study. Between the final and follow-up analyses, 1 patient was found to have an invalid ICF and was not included in the follow-up analysis.
Measure: Number; unit: First events per person-year
Arm/Group | MAGE-A3 Group | Placebo Group | GS+ Mage-A3 Sub-Group | GS+ Placebo Sub-Group | GS- Mage-A3 Sub-Group | GS- Placebo Sub-Group
Number analyzed (Participants) | 892 | 452 | 200 | 116 | 255 | 126
First events per person-year | 0.366 | 0.345 | 0.345 | 0.335 | 0.316 | 0.319
Statistical Analysis 1: Comparison: MAGE-A3 Group vs Placebo Group; At Follow-up analysis (up to Year 5); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.7534, Regression, Cox; Hazard Ratio (HR) = 1.023, 95% CI 2-sided [0.890 to 1.175]
Statistical Analysis 2: Comparison: GS+ Mage-A3 Sub-Group vs GS+ Placebo Sub-Group; At Follow-up analysis (up to Year 5); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.5385, Regression, Cox; Hazard Ratio (HR) = 1.094, 95% CI 2-sided [0.821 to 1.457]
Statistical Analysis 3: Comparison: GS- Mage-A3 Sub-Group vs GS- Placebo Sub-Group; At Follow-up analysis (up to Year 5); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 3]; p = 0.5419, Regression, Cox; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.698 to 1.207]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time to event from randomization to the date of death, irrespective of the cause of death. OS was expressed as the person-year rate i.e. the number of patients with death (n) over the sum of the follow-up periods in years (T). Patients alive at the time of the analysis were censored on the date last known to be alive.
Time Frame: At Final analysis (Month 30 = Year 2.5) and at follow-up analysis (up to Year 5)
Population: as for outcome 2
Measure: Number; unit: Events per person-year
Groups:
- GS+ Mage-A3 Sub-Group: Subset of patients with the pre-specified gene signature, receiving the MAGE-A3 ASCI product. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of ASCI product at 3-week intervals, followed by 8 doses of ASCI product at 12-week intervals.
- GS- Mage-A3 Sub-Group: Subset of patients without the pre-specified gene signature, receiving the MAGE-A3 ASCI product. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening. Study products were administered as intramuscular (IM) injections in the deltoid or the lateral region of the thigh (not in anatomical regions where lymph nodes had been excised): 5 doses of ASCI product at 3-week intervals, followed by 8 doses of ASCI product at 12-week intervals.
Arm/Group | MAGE-A3 Group | Placebo Group | GS+ Mage-A3 Sub-Group | GS+ Placebo Sub-Group | GS- Mage-A3 Sub-Group | GS- Placebo Sub-Group
Number analyzed (Participants) | 893 | 452 | 200 | 116 | 255 | 126
Events per person-year
  OS, Final analysis | 0.177 | 0.165 | 0.172 | 0.188 | 0.165 | 0.151
  OS, Follow-up analysis: number analyzed (Participants) | 892 | 452 | 200 | 116 | 255 | 126
  OS, Follow-up analysis | 0.146 | 0.140 | 0.146 | 0.153 | 0.132 | 0.120

4. Secondary Outcome: Disease-free Specific Survival (DFSS)
Description: Disease Free Specific Survival (DFSS) was defined as the time to event from randomization to the date of first recurrence of disease or date of death due to melanoma (cause as assessed by investigator), whichever occurred first. DFSS was expressed as the person-year rate i.e. the number of patients with at least one event (n) over the sum of the follow-up periods in years (T), until the first occurrence of a recurrence/death. Patients who died due to a cause other than the disease under study and patients alive at the time of analysis were censored on the date of last assessment (visit or tumor assessment).
Time Frame: At Final analysis (Month 30 = Year 2.5)
Population: as for outcome 1
Measure: Number; unit: First events per person-year
Arm/Group | MAGE-A3 Group | Placebo Group | GS+ Mage-A3 Sub-Group | GS- Mage-A3 Sub-Group | GS+ Placebo Sub-Group | GS- Placebo Sub-Group
Number analyzed (Participants) | 893 | 452 | 200 | 116 | 255 | 126
First events per person-year | 0.499 | 0.478 | 0.500 | 0.460 | 0.434 | 0.442

5. Secondary Outcome: Distant Metastasis-free Survival (DMFS)
Description: Distant Metastasis Free Survival (DMFS) was defined as the time to event from randomization to the date of first distant metastasis or date of death, whichever occurred first. DMFS was expressed as the person-year rate i.e. the number of patients with at least one event (n) over the sum of the follow-up periods in years (T), until the first occurrence of distant metastasis/death. Patients alive and without distant metastases were censored at the date of last assessment (visit or tumor assessment, or date of last tumor assessment as documented during the yearly contact follow-up period).
Time Frame: At Final analysis (Month 30 = Year 2.5)
Population: as for outcome 1
Measure: Number; unit: First events per person-year
Arm/Group | MAGE-A3 Group | Placebo Group | GS+ Mage-A3 Sub-Group | GS+ Placebo Sub-Group | GS- Mage-A3 Sub-Group | GS- Placebo Sub-Group
Number analyzed (Participants) | 893 | 452 | 200 | 116 | 255 | 126
First events per person-year | 0.387 | 0.342 | 0.388 | 0.337 | 0.334 | 0.307

6. Secondary Outcome: Health-related Quality of Life
Description: The assessment of health-related quality of life was restricted to patients who consented to study participation after Protocol Amendment 1 became effective at their study site, and for whom a validated version of the Euro Quality of Life-5D (EQ-5D) questionnaire was available in their native language. The EQ-5D comprises a 5-dimensional descriptive system (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), where each item has 3 levels and together they define 243 possible health states. For each health state, a value (utility) was determined by using an additive algorithm. These utility scores were calculated for each patient at each timepoint at which an EQ-5D questionnaire was completed. The score had a maximum value of 1.0 corresponding to full health level, while lower scores, down to a minimum value of 0.0 reflected degradation in the health-related quality of life.
Time Frame: At Weeks 0, 6, 12 [on the day of and the day after treatment administration (TA)], at Month 6, 9, 12, 24, at the Concluding visit (Month 30) + 6 months and +12 Months and at disease recurrence
Population: The analysis was performed on subjects with valid EQ-5D data from the Total Treated population - as randomized, which included patients in the treatment groups as allocated by the randomization system at the start of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 245 | 118
Units on a scale
  EQ-5D, Week 0 (day of TA) | 0.842 (0.182) | 0.861 (0.159)
  EQ-5D, Week 0 (day after TA): number analyzed (Participants) | 195 | 94
  EQ-5D, Week 0 (day after TA) | 0.773 (0.182) | 0.873 (0.141)
  EQ-5D, Week 6 (day of TA): number analyzed (Participants) | 234 | 118
  EQ-5D, Week 6 (day of TA) | 0.853 (0.183) | 0.865 (0.173)
  EQ-5D, Week 6 (day after TA): number analyzed (Participants) | 198 | 96
  EQ-5D, Week 6 (day after TA) | 0.722 (0.245) | 0.867 (0.174)
  EQ-5D, Week 12 (day of TA): number analyzed (Participants) | 193 | 96
  EQ-5D, Week 12 (day of TA) | 0.873 (0.158) | 0.887 (0.138)
  EQ-5D, Week 12 (day after TA): number analyzed (Participants) | 162 | 77
  EQ-5D, Week 12 (day after TA) | 0.788 (0.170) | 0.888 (0.126)
  EQ-5D, Month 6: number analyzed (Participants) | 144 | 75
  EQ-5D, Month 6 | 0.879 (0.146) | 0.900 (0.156)
  EQ-5D, Month 9: number analyzed (Participants) | 130 | 77
  EQ-5D, Month 9 | 0.891 (0.134) | 0.876 (0.194)
  EQ-5D, Month 12: number analyzed (Participants) | 113 | 67
  EQ-5D, Month 12 | 0.891 (0.157) | 0.899 (0.149)
  EQ-5D, Month 24: number analyzed (Participants) | 62 | 36
  EQ-5D, Month 24 | 0.894 (0.132) | 0.881 (0.150)
  EQ-5D, Month 30 + 6 months: number analyzed (Participants) | 1 | 2
  EQ-5D, Month 30 + 6 months | 0.727 (0.000) | 0.568 (0.074)
  EQ-5D, Month 30 + 12 months: number analyzed (Participants) | 30 | 10
  EQ-5D, Month 30 + 12 months | 0.791 (0.264) | 0.648 (0.344)
  EQ-5D, Disease recurrence: number analyzed (Participants) | 76 | 35
  EQ-5D, Disease recurrence | 0.752 (0.261) | 0.815 (0.197)

7. Secondary Outcome: Number of Subjects With Anti-MAGE-A3 Antibody Concentrations Above the Cut-off Value
Description: The cut-off value was 27 Enzyme-Linked Immunosorbent Assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Weeks 0, 6, 12, 36, 48 72, 120 (Concluding visit) and at Week 120 + 6 months
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all eligible subjects who have received at least the first 4 MAGE-A3 ASCI study treatment doses and have provided a result for immunogenicity measurement within the time schedule for study product administration and blood sample draw.
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 629 | 316
Participants
  Anti-MAGE-A3, Week 0 | 25 | 19
  Anti-MAGE-A3, Week 6: number analyzed (Participants) | 482 | 271
  Anti-MAGE-A3, Week 6 | 478 | 22
  Anti-MAGE-A3, Week 12: number analyzed (Participants) | 425 | 230
  Anti-MAGE-A3, Week 12 | 424 | 13
  Anti-MAGE-A3, Week 36: number analyzed (Participants) | 259 | 131
  Anti-MAGE-A3, Week 36 | 259 | 6
  Anti-MAGE-A3, Week 48: number analyzed (Participants) | 224 | 113
  Anti-MAGE-A3, Week 48 | 224 | 5
  Anti-MAGE-A3, Week 72: number analyzed (Participants) | 178 | 85
  Anti-MAGE-A3, Week 72 | 178 | 4
  Anti-MAGE-A3, Week 120: number analyzed (Participants) | 257 | 140
  Anti-MAGE-A3, Week 120 | 257 | 10
  Anti-MAGE-A3, Week 120+6 months: number analyzed (Participants) | 70 | 36
  Anti-MAGE-A3, Week 120+6 months | 70 | 1

8. Secondary Outcome: Anti-MAGE-A3 Antibody Geometric Mean Concentrations
Description: Anti-MAGE-A3 antibody concentrations were presented as geometric mean concentrations (GMC) and expressed in EL.U/mL.
Time Frame: At Weeks 0, 6, 12, 36, 48 72, 120 (Concluding visit) and at Month 120 + 6 months
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 629 | 316
EL.U/mL
  Anti-MAGE-A3, Week 0 | 11.0 [10.6 to 11.4] | 11.4 [10.7 to 12.1]
  Anti-MAGE-A3, Week 6: number analyzed (Participants) | 482 | 271
  Anti-MAGE-A3, Week 6 | 1451.6 [1290.9 to 1632.3] | 11.9 [11.0 to 12.9]
  Anti-MAGE-A3, Week 12: number analyzed (Participants) | 425 | 230
  Anti-MAGE-A3, Week 12 | 4031.6 [3738.7 to 4347.4] | 11.3 [10.6 to 12.1]
  Anti-MAGE-A3, Week 36: number analyzed (Participants) | 259 | 131
  Anti-MAGE-A3, Week 36 | 2189.6 [2000.4 to 2396.7] | 11.4 [10.4 to 12.4]
  Anti-MAGE-A3, Week 48: number analyzed (Participants) | 224 | 113
  Anti-MAGE-A3, Week 48 | 2243.4 [2034.4 to 2473.8] | 11.3 [10.2 to 12.6]
  Anti-MAGE-A3, Week 72: number analyzed (Participants) | 178 | 85
  Anti-MAGE-A3, Week 72 | 2489.4 [2221.8 to 2789.4] | 11.2 [10.0 to 12.5]
  Anti-MAGE-A3, Week 120: number analyzed (Participants) | 257 | 140
  Anti-MAGE-A3, Week 120 | 3109.7 [2827.4 to 3420.2] | 12.7 [10.9 to 14.8]
  Anti-MAGE-A3, Week 120+6 months: number analyzed (Participants) | 70 | 36
  Anti-MAGE-A3, Week 120+6 months | 1293.4 [1056.3 to 1583.7] | 10.8 [9.9 to 11.8]

9. Secondary Outcome: Number of Subjects With Anti-MAGE-A3 Antibody Response
Description: Treatment response defined as: - For initially seronegative patients: post-treatment antibody concentration ≥ 27 EL.U/mL; - For initially seropositive patients: post-treatment antibody concentration ≥ 2 fold the pre-treatment antibody concentration.
Time Frame: At Weeks 6, 12, 36, 48 72, 120 (Concluding visit) and at Month 120 + 6 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 482 | 271
Participants
  Anti-MAGE-A3, Week 6 | 476 | 9
  Anti-MAGE-A3, Week 12: number analyzed (Participants) | 425 | 230
  Anti-MAGE-A3, Week 12 | 424 | 4
  Anti-MAGE-A3, Week 36: number analyzed (Participants) | 259 | 131
  Anti-MAGE-A3, Week 36 | 259 | 2
  Anti-MAGE-A3, Week 48: number analyzed (Participants) | 224 | 113
  Anti-MAGE-A3, Week 48 | 224 | 2
  Anti-MAGE-A3, Week 72: number analyzed (Participants) | 178 | 85
  Anti-MAGE-A3, Week 72 | 178 | 2
  Anti-MAGE-A3, Week 120: number analyzed (Participants) | 257 | 140
  Anti-MAGE-A3, Week 120 | 257 | 6
  Anti-MAGE-A3, Week 120+6 months: number analyzed (Participants) | 70 | 36
  Anti-MAGE-A3, Week 120+6 months | 70 | 1

10. Secondary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Parameters
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: alanine aminotransferase [ALT], asparatate aminostransferase [AST], alkaline phoshatase [AP], bilirubin [BIL], creatinine [CREA], hemoglobin [HGB], leukocytes [LEU], lymphopenia [LYMPH], neutrophils [NEU], platelets [PLA]. Parameter grades (Grade [G] 0, 1, 2, 3, 4, Unknown) were compared to each baseline parameter grade (G Unknown, 0, 1, 2, 3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 of August 9, 2006.
Time Frame: Within the 31-day (Days 0-30) post-treatment period
Population: The analysis was performed on the Total Treated population - as treated, which included patients in the treatment group as per treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 894 | 450
Participants
  ALT, Unknown - G0 | 3 | 2
  ALT, Unknown - G1 | 1 | 0
  ALT, Unknown - G2 | 0 | 0
  ALT, Unknown - G3 | 0 | 0
  ALT, Unknown - G4 | 0 | 0
  ALT, Unknown - Unknown | 2 | 0
  ALT, G0 - G0 | 625 | 337
  ALT, G0 - G1 | 98 | 30
  ALT, G0 - G2 | 10 | 4
  ALT, G0 - G3 | 3 | 4
  ALT, G0 - G4 | 0 | 0
  ALT, G0 - Unknown | 36 | 18
  ALT, G1 - G0 | 45 | 22
  ALT, G1 - G1 | 49 | 25
  ALT, G1 - G2 | 14 | 4
  ALT, G1 - G3 | 1 | 2
  ALT, G1 - G4 | 0 | 0
  ALT, G1 - Unknown | 2 | 1
  ALT, G2 - G0 | 1 | 1
  ALT, G2 - G1 | 2 | 0
  ALT, G2 - G2 | 1 | 0
  ALT, G2 - G3 | 0 | 0
  ALT, G2 - G4 | 0 | 0
  ALT, G2 - Unknown | 0 | 0
  ALT, G3 - G0 | 0 | 0
  ALT, G3 - G1 | 0 | 0
  ALT, G3 - G2 | 0 | 0
  ALT, G3 - G3 | 0 | 0
  ALT, G3 - G4 | 0 | 0
  ALT, G3 - Unknown | 1 | 0
  ALT, Total - G0 | 674 | 362
  ALT, Total - G1 | 150 | 55
  ALT, Total - G2 | 25 | 8
  ALT, Total - G3 | 4 | 6
  ALT, Total - G4 | 0 | 0
  ALT, Total - Unknown | 41 | 19
  AST, Unknown - G0 | 3 | 3
  AST, Unknown - G1 | 1 | 0
  AST, Unknown - G2 | 0 | 0
  AST, Unknown - G3 | 0 | 0
  AST, Unknown - G4 | 0 | 0
  AST, Unknown - Unknown | 3 | 0
  AST, G0 - G0 | 701 | 356
  AST, G0 - G1 | 88 | 37
  AST, G0 - G2 | 5 | 3
  AST, G0 - G3 | 3 | 4
  AST, G0 - G4 | 0 | 0
  AST, G0 - Unknown | 40 | 19
  AST, G1 - G0 | 24 | 15
  AST, G1 - G1 | 18 | 11
  AST, G1 - G2 | 3 | 1
  AST, G1 - G3 | 2 | 0
  AST, G1 - G4 | 0 | 0
  AST, G1 - Unknown | 1 | 1
  AST, G2 - G0 | 0 | 0
  AST, G2 - G1 | 0 | 0
  AST, G2 - G2 | 1 | 0
  AST, G2 - G3 | 0 | 0
  AST, G2 - G4 | 0 | 0
  AST, G2 - Unknown | 1 | 0
  AST, Total - G0 | 728 | 374
  AST, Total - G1 | 107 | 48
  AST, Total - G2 | 9 | 4
  AST, Total - G3 | 5 | 4
  AST, Total - G4 | 0 | 0
  AST, Total - Unknown | 45 | 20
  AP, Unknown - G0 | 9 | 6
  AP, Unknown - G1 | 0 | 1
  AP, Unknown - G2 | 1 | 0
  AP, Unknown - G3 | 0 | 0
  AP, Unknown - G4 | 0 | 0
  AP, Unknown - Unknown | 2 | 0
  AP, G0 - G0 | 749 | 378
  AP, G0 - G1 | 56 | 18
  AP, G0 - G2 | 3 | 4
  AP, G0 - G3 | 2 | 1
  AP, G0 - G4 | 0 | 0
  AP, G0 - Unknown | 38 | 18
  AP, G1 - G0 | 18 | 13
  AP, G1 - G1 | 14 | 9
  AP, G1 - G2 | 0 | 0
  AP, G1 - G3 | 0 | 0
  AP, G1 - G4 | 0 | 0
  AP, G1 - Unknown | 2 | 2
  AP, Total - G0 | 776 | 397
  AP, Total - G1 | 70 | 28
  AP, Total - G2 | 4 | 4
  AP, Total - G3 | 2 | 1
  AP, Total - G4 | 0 | 0
  AP, Total - Unknown | 42 | 20
  BIL, Unknown - G0 | 7 | 5
  BIL, Unknown - G1 | 1 | 0
  BIL, Unknown - G2 | 0 | 0
  BIL, Unknown - G3 | 0 | 0
  BIL, Unknown - G4 | 0 | 0
  BIL, Unknown - Unknown | 1 | 1
  BIL, G0 - G0 | 771 | 383
  BIL, G0 - G1 | 33 | 21
  BIL, G0 - G2 | 3 | 2
  BIL, G0 - G3 | 0 | 1
  BIL, G0 - G4 | 0 | 0
  BIL,G 0 - Unknown | 44 | 19
  BIL, G1 -G 0 | 11 | 3
  BIL, G1 - G1 | 10 | 5
  BIL, G1 -G 2 | 9 | 4
  BIL, G1 - G3 | 0 | 0
  BIL, G1 - G4 | 0 | 0
  BIL, G1 - Unknown | 3 | 2
  BIL, G2 - G0 | 0 | 0
  BIL, G2 - G1 | 0 | 2
  BIL, G2 - G2 | 0 | 2
  BIL, G2 - G3 | 0 | 0
  BIL, G2 - G4 | 0 | 0
  BIL, G2 - Unknown | 1 | 0
  BIL, Total - G0 | 789 | 391
  BIL, Total - G1 | 44 | 28
  BIL, Total - G2 | 12 | 8
  BIL, Total - G3 | 0 | 1
  BIL, Total - G4 | 0 | 0
  BIL, Total - Unknown | 49 | 22
  CREA, Unknown - G0 | 2 | 1
  CREA, Unknown - G1 | 0 | 0
  CREA, Unknown - G2 | 0 | 0
  CREA, Unknown - G3 | 0 | 0
  CREA, Unknown - G4 | 0 | 0
  CREA, Unknown - Unknown | 1 | 0
  CREA, G0 - G0 | 789 | 391
  CREA, G0 - G1 | 31 | 19
  CREA, G0 - G2 | 0 | 1
  CREA, G0 - G3 | 0 | 1
  CREA, G0 - G4 | 0 | 0
  CREA, G0 - Unknown | 36 | 19
  CREA, G1 - G0 | 8 | 6
  CREA, G1 - G1 | 19 | 12
  CREA, G1 - G2 | 3 | 0
  CREA, G1 - G3 | 0 | 0
  CREA, G1 - G4 | 0 | 0
  CREA, G1 - Unknown | 4 | 0
  CREA, G2 - G0 | 0 | 0
  CREA, G2 - G1 | 0 | 0
  CREA, G2 - G2 | 1 | 0
  CREA, G2 - G3 | 0 | 0
  CREA, G2 - G4 | 0 | 0
  CREA, G2 - Unknown | 0 | 0
  CREA, Total - G0 | 799 | 398
  CREA, Total - G1 | 50 | 31
  CREA, Total - G2 | 4 | 1
  CREA, Total - G3 | 0 | 1
  CREA, Total - G4 | 0 | 0
  CREA, Total - Unknown | 41 | 19
  HGB, Unknown - G0 | 2 | 1
  HGB, Unknown - G1 | 1 | 0
  HGB, Unknown - G2 | 0 | 0
  HGB, Unknown - G3 | 0 | 0
  HGB, Unknown - G4 | 0 | 0
  HGB, Unknown - Unknown | 0 | 0
  HGB, G0 - G0 | 636 | 326
  HGB, G0 - G1 | 78 | 28
  HGB, G0 - G2 | 7 | 3
  HGB, G0 - G3 | 2 | 1
  HGB, G0 - G4 | 0 | 0
  HGB, G0 - Unknown | 35 | 17
  HGB, G1 - G0 | 39 | 27
  HGB, G1 - G1 | 77 | 41
  HGB, G1 - G2 | 7 | 2
  HGB, G1 - G3 | 1 | 0
  HGB, G1 - G4 | 1 | 0
  HGB, G1 - Unknown | 4 | 3
  HGB, G2 - G0 | 1 | 1
  HGB, G2 - G1 | 1 | 0
  HGB, G2 - G2 | 2 | 0
  HGB, G2 - G3 | 0 | 0
  HGB, G2 - G4 | 0 | 0
  HGB, G2 - Unknown | 0 | 0
  HGB, Total - G0 | 678 | 355
  HGB, Total - G1 | 157 | 69
  HGB, Total - G2 | 16 | 5
  HGB, Total - G3 | 3 | 1
  HGB, Total - G4 | 1 | 0
  HGB, Total - Unknown | 39 | 20
  LEU, Unknown - G0 | 2 | 1
  LEU, Unknown - G1 | 1 | 0
  LEU, Unknown - G2 | 0 | 0
  LEU, Unknown - G3 | 0 | 0
  LEU, Unknown - G4 | 0 | 0
  LEU, Unknown - Unknown | 0 | 0
  LEU, G0 - G0 | 762 | 382
  LEU, G0 - G1 | 53 | 31
  LEU, G0 - G2 | 4 | 2
  LEU, G0 - G3 | 0 | 0
  LEU, G0 - G4 | 2 | 0
  LEU, G0 - Unknown | 39 | 18
  LEU, G1 - G0 | 13 | 8
  LEU, G1 - G1 | 15 | 6
  LEU, G1 - G2 | 1 | 1
  LEU, G1 - G3 | 0 | 0
  LEU, G1 - G4 | 0 | 0
  LEU, G1 - Unknown | 0 | 1
  LEU, G2 - G0 | 0 | 0
  LEU, G2 - G1 | 1 | 0
  LEU, G2 - G2 | 0 | 0
  LEU, G2 - G3 | 1 | 0
  LEU, G2 - G4 | 0 | 0
  LEU, G2 - Unknown | 0 | 0
  LEU, Total - G0 | 777 | 391
  LEU, Total - G1 | 70 | 37
  LEU, Total - G2 | 5 | 3
  LEU, Total - G3 | 1 | 0
  LEU, Total - G4 | 2 | 0
  LEU, Total - Unknown | 39 | 19
  LYMPH, Unknown - G0 | 8 | 1
  LYMPH, Unknown - G1 | 2 | 2
  LYMPH, Unknown - G2 | 0 | 0
  LYMPH, Unknown - G3 | 0 | 0
  LYMPH, Unknown - G4 | 0 | 0
  LYMPH, Unknown - Unknown | 0 | 0
  LYMPH, G0 - G0 | 633 | 303
  LYMPH, G0 - G1 | 93 | 57
  LYMPH, G0 - G2 | 17 | 8
  LYMPH, G0 - G3 | 4 | 0
  LYMPH, G0 - G4 | 0 | 0
  LYMPH, G0 - Unknown | 38 | 22
  LYMPH, G1 - G0 | 29 | 9
  LYMPH, G1 - G1 | 49 | 37
  LYMPH, G1 - G2 | 4 | 6
  LYMPH, G1 - G3 | 4 | 0
  LYMPH, G1 - G4 | 0 | 0
  LYMPH, G1 - Unknown | 4 | 0
  LYMPH, G2 - G0 | 1 | 1
  LYMPH, G2 - G1 | 4 | 1
  LYMPH, G2 - G2 | 2 | 2
  LYMPH, G2 - G3 | 2 | 0
  LYMPH, G2 - G4 | 0 | 0
  LYMPH, G2 - Unknown | 0 | 0
  LYMPH, G3 - G0 | 0 | 0
  LYMPH, G3 - G1 | 0 | 1
  LYMPH, G3 - G2 | 0 | 0
  LYMPH, G3 - G3 | 0 | 0
  LYMPH, G3 - G4 | 0 | 0
  LYMPH, G3 - Unknown | 0 | 0
  LYMPH, Total - G0 | 671 | 314
  LYMPH, Total - G1 | 148 | 98
  LYMPH, Total - G2 | 23 | 16
  LYMPH, Total - G3 | 10 | 0
  LYMPH, Total - G4 | 0 | 0
  LYMPH, Total - Unknown | 42 | 22
  NEU, Unknown - G0 | 6 | 1
  NEU, Unknown - G1 | 0 | 1
  NEU, Unknown - G2 | 0 | 0
  NEU, Unknown - G3 | 0 | 0
  NEU, Unknown - G4 | 0 | 0
  NEU, Unknown - Unknown | 0 | 0
  NEU, G0 - G0 | 781 | 393
  NEU, G0 - G1 | 39 | 16
  NEU, G0 - G2 | 9 | 2
  NEU, G0 - G3 | 0 | 0
  NEU, G0 - G4 | 1 | 0
  NEU, G0 - Unknown | 43 | 22
  NEU, G1 - G0 | 7 | 10
  NEU, G1 - G1 | 6 | 3
  NEU, G1 - G2 | 1 | 2
  NEU, G1 - G3 | 0 | 0
  NEU, G1 - G4 | 0 | 0
  NEU, G1 - Unknown | 0 | 0
  NEU, G2 - G0 | 0 | 0
  NEU, G2 - G1 | 1 | 0
  NEU, G2 - G2 | 0 | 0
  NEU, G2 - G3 | 0 | 0
  NEU, G2 - G4 | 0 | 0
  NEU, G2 - Unknown | 0 | 0
  NEU, Total - G0 | 794 | 404
  NEU, Total - G1 | 46 | 20
  NEU, Total - G2 | 10 | 4
  NEU, Total - G3 | 0 | 0
  NEU, Total - G4 | 1 | 0
  NEU, Total - Unknown | 43 | 22
  PLA, Unknown - G0 | 4 | 1
  PLA, Unknown - G1 | 0 | 0
  PLA, Unknown - G2 | 0 | 0
  PLA, Unknown - G3 | 0 | 0
  PLA, Unknown - G4 | 0 | 0
  PLA, Unknown - Unknown | 0 | 0
  PLA, G0 - G0 | 796 | 390
  PLA, G0 - G1 | 34 | 25
  PLA, G0 - G2 | 0 | 1
  PLA, G0 - G3 | 0 | 0
  PLA, G0 - G4 | 1 | 3
  PLA, G0 - Unknown | 36 | 17
  PLA, G1 - G0 | 4 | 1
  PLA, G1 - G1 | 15 | 10
  PLA, G1 - G2 | 1 | 0
  PLA, G1 - G3 | 0 | 0
  PLA, G1 - G4 | 0 | 0
  PLA, G1 - Unknown | 3 | 2
  PLA, Total - G0 | 804 | 392
  PLA, Total - G1 | 49 | 35
  PLA, Total - G2 | 1 | 1
  PLA, Total - G3 | 0 | 0
  PLA, Total - G4 | 1 | 3
  PLA, Total - Unknown | 39 | 19

11. Secondary Outcome: Number of Subjects With Any Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 31-day (Days 0-30) follow-up period after treatment
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 895 | 450
Participants | 822 | 333

12. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to study end (up to 5 years)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 895 | 450
Participants | 129 | 64

13. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 0 up to study end (up to 5 years)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | MAGE-A3 Group | Placebo Group
Number analyzed (Participants) | 895 | 450
Participants | 33 | 23

ADVERSE EVENTS:
Time Frame: Adverse events (AEs): Within the 31-day (Days 0-30) follow-up period after treatment. Serious Adverse Events: from Day 0 up to study end (up to 5 years).
Arm/Group | MAGE-A3 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 5/895 | 1/450
Serious Adverse Events (participants affected / at risk) | 129/895 | 64/450
Other Adverse Events (participants affected / at risk) | 819/895 | 327/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAGE-A3 Group (N=895) | Placebo Group (N=450)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Polyglandular autoimmune syndrome type ii (Endocrine disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinal vascular thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 5 (5)
Cellulitis enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 7 (9) | 5 (5)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
H1n1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph node abscess (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 2 (2) | 0 (0)
Prostatitis escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electric shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (34) | 13 (14)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 3 (3)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant melanoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (9) | 3 (3)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Meningism (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (2)
Bladder neck sclerosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic elastosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAGE-A3 Group (N=895) | Placebo Group (N=450)
Diarrhoea (Gastrointestinal disorders) | 46 (61) | 19 (26)
Nausea (Gastrointestinal disorders) | 123 (266) | 32 (43)
Asthenia (General disorders) | 149 (354) | 46 (68)
Chills (General disorders) | 179 (432) | 15 (23)
Fatigue (General disorders) | 210 (490) | 63 (116)
Influenza like illness (General disorders) | 261 (902) | 30 (46)
Injection site erythema (General disorders) | 90 (241) | 3 (3)
Injection site oedema (General disorders) | 48 (134) | 3 (5)
Injection site pain (General disorders) | 325 (1057) | 22 (37)
Injection site reaction (General disorders) | 160 (500) | 6 (9)
Pain (General disorders) | 191 (480) | 19 (26)
Pyrexia (General disorders) | 380 (1240) | 35 (44)
Arthralgia (Musculoskeletal and connective tissue disorders) | 84 (165) | 31 (43)
Myalgia (Musculoskeletal and connective tissue disorders) | 188 (456) | 23 (39)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 115 (207) | 26 (28)
Headache (Nervous system disorders) | 205 (550) | 55 (128)
Erythema (Skin and subcutaneous tissue disorders) | 138 (297) | 10 (10)

LIMITATIONS AND CAVEATS:
The study was terminated early on 08 Sep 2015 following assessment of the two co-primary endpoints showed the lack of efficacy of the study product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.